CLINICAL TRIAL: NCT06524895
Title: Pilot Study of Medical Reiki for Women Undergoing Surgery for Breast Cancer: Impact on Quality of Life, Medical Recovery Metrics, and Cortisol
Brief Title: Reiki Breast Surgery QOL Project for Women Undergoing Breast Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Medical Reiki Works, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-14017
Record Dates: First submitted 2024-07-25; First posted 2024-07-29 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Reiki
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Consented participants will be allocated in a 1:1 ratio between the Reiki and the Sham Reiki arms. Participants will be assigned to the intervention arms using a permuted block randomized design. Blocks of two (75%) and four (25%) will be used to randomize patients.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to intervention assignment so in every other aspect aside from the "energy healing", Sham practitioners should resemble the Reiki healers, and will be stratified by surgery type. Clinical staff who take objective recovery metrics will be blinded to the intervention and control arm status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Medical Reiki (Active Comparator): The energy medicine will be delivered to the study participant immediately pre-op. The Reiki practitioner will hold the participant's hand for 10 minutes. This will be followed by touching the participant's upper arm along with shoulder for 20 minutes. Clinical staff will ask standard questions to assess mood while receiving the energy medicine. Because this is a medical study, the practitioner will mainly be silent for the 30 minute session.
  Interventions: Other: Medical Reiki
- Group B- Sham Reiki (Sham Comparator): Patients will be recruited to receive "Sham" Reiki before surgery. The non-Reiki healer will hold the participant's hand for 10 minutes. This will be followed by touching the participant's upper arm along with shoulder for 20 minutes. Clinical staff will ask standard questions to assess mood while receiving the energy medicine. Because this is a medical study, the non-Reiki healer will mainly be silent for the 30 minute session.
  Interventions: Other: Sham Reiki

INTERVENTIONS:
Other: Medical Reiki — Reiki is a form of energy therapy involving the facilitation of healing through the manipulation of biofields utilizing light touch. It is a process of targeting the energy fields around the patient's body is believed to stimulate the patient's natural ability to heal itself.
  Arms: Group A- Medical Reiki
Other: Sham Reiki — Sham Reiki involves a non-Reiki healer who mimics the treatment of a Reiki healer. Sham Reiki providers will be medical students who are not interested and without prior knowledge or experience with Reiki Medicine.The medical students will not have any prior experience in Reiki healing or associated energy healing modalities. It is better for this project if the medical student has no interest so there is true placebo effect being monitored.
  Arms: Group B- Sham Reiki

SUMMARY:
This pilot study will examine the impact of pre-operative Medical Reiki© on the psychosocial well-being and recovery of underserved women undergoing breast cancer surgery.

DETAILED DESCRIPTION:
Reiki is a form of energy therapy involving the facilitation of healing through the manipulation of biofields utilizing light touch. Practitioners lightly place their hands directly on or above the patient's body to transmit energy from the practitioner to the recipient. This process of targeting the energy fields around the patient's body is believed to stimulate the patient's natural ability to heal itself. Reiki is a safe treatment modality that emphasizes spirituality in healing and wellness whose origins are rooted in ancient Tibetan traditions. The prevalence of integrating complementary therapies such as Reiki into mainstream medical practices is demonstrated by the number of hospitals that make use of these therapies to help alleviate, for example, the fatigue, pain, anxiety, and diminished quality of life experienced by cancer patients and those with other illnesses. Reiki in particular, has become more widespread in cancer centers because of its potential to reduce cancer-related symptoms and enhanced wellness without posing harm to patients.

A pilot double-blind randomized-controlled design will be used to engage 32 women in a pre-operative Reiki intervention designed by Raven Keyes called Medical Reiki© with a follow-up of two months. Women diagnosed with stage I-III breast cancer undergoing mastectomy for their treatment will be recruited to study within two weeks of surgery. Patients will be recruited to receive Medical Reiki© vs Sham Reiki (attention control) before surgery, with medical and psychosocial outcomes assessment conducted at three time points: -T0 - Baseline/pre-surgery; T1 (1-month); T2 (2 months). These assessments will either be self-administered or administered via telephone by the research team. The study The study will aim to determine the feasibility of offering Medical Reiki to breast cancer patients immediately prior to breast surgery; the impact of pre-operative Medical Reiki© vs Sham Reiki on post-operative recovery at the identified timepoints based on the specified measures of Subjective QoL metrics and objective recovery metrics.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-99
* Breast Cancer Diagnosis Stage 0-III
* Undergoing unilateral or bilateral mastectomy (with or without reconstruction) within 2 weeks of recruitment
* English Speaking
* From within 50 miles of Bronx County, NY

Exclusion Criteria:

* Current, uncontrolled psychiatric co-morbidities
* Pregnant women

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility based on Number Screened for Inclusion | 2 months
  The total number of patients screened for inclusion will be summarized and reported.
Feasibility - Percentage of Patients who met Inclusion Criteria | 2 months
  The number/percentage of patients who met inclusion criteria will be summarized and reported.
Feasibility - Percentage of Patients who Assented for Informed Consent | 2 months
  The number/percentage of patients who assented for Informed Consent will be summarized and reported.
Feasibility - Percentage of Patients who Completed the Informed Consent Procedure | 2 months
  The number/percentage of patients who completed the Informed Consent Procedure will be summarized and reported.
Feasibility - Percentage of Patients who Agreed and Refused to Participate | 2 months
  The number/percentage of patients who agreed/refused to Participate will be summarized and reported.
Feasibility - Percentage of Patients who Completed Baseline Assessments | 2 months
  The number/percentage of patients who completed baseline assessments will be summarized and reported.
Feasibility - Percentage of Patients who were Randomly Allocated as per allocation list to Treatment Arm | 2 months
  The number/percentage of patients who who were Randomly Allocated as per allocation list to Treatment Arm will be summarized and reported.
Feasibility - Percentage of Patients who Received Intended Intervention | 2 months
  The number/percentage of patients who received the intended intervention will be summarized and reported.
Feasibility - Percentage of Patients who Dropped out during Follow-up Visits | 2 months
  The number/percentage of patients who dropped out during follow-up Visits will be summarized and reported.
Feasibility - Percentage of Patients who Completed all End Line Assessments | 2 months
  The number/percentage of patients who completed all end Line assessments will be summarized and reported.
Feasibility - Percentage of Patients who were Unmasked during End Line Assessments | 2 months
  The number/percentage of patients who were Unmasked during End Line Assessments will be summarized and reported.
Feasibility - Retention Rate | 2 months post-operatively
  Feasibility will be assessed based on retention of study patients in the study arms. For this study retention rate will be determined per study arm and will be equal to the ratio (in percentage) of the number of patients who completed all study activities at two months to the number of patients assigned to that study arm. For this study a retention rate of 80% is targeted.
Provider Fidelity | Immediately after intervention (before surgery), up to 1 hour
  Provider fidelity will be assessed based upon responses to a Reiki Fidelity Provider Survey administered immediately after the intervention session. The survey consists of 11 questions (including one question which contains three sub-questions). For purposes of assessing Provider Fidelity only the first three questions on the survey are scored. For these three questions, providers are asked to identify a score on an 11-point Likert scale ranging from 0 (either "Not at all" or "Uncomfortable") to 10 (either "Completely" or "Very Comfortable") as to the conduct of the intervention, the degree of comfort they felt, and the degree of comfort providers perceived that their patients felt, during the session, for an overall possible scoring range of 0-30. Higher scores associated with and increased level of provider fidelity. Overall scores will be summarized at each time point using basic descriptive statistics.
Patient Fidelity | Immediately after intervention (before surgery), up to 1 hour
  Patient fidelity will be assessed based upon responses to a Reiki Fidelity Patient Survey administered immediately following the intervention session. The survey consists of 8 questions; however, for purposes of assessing Patient Fidelity only questions 1, 2, 6, and 7 on the survey are scored. For these four questions, patients are asked to identify a score on an 11-point Likert scale ranging from 0 (either "Very Negative", "Uncomfortable", or "Not at all") to 10 (either "Very Positive", "Very Comfortable", or "Very Much") as to their experience with the intervention, their level of comfort with the intervention and their expectations as to the impact on physical and emotional recovery derived from the intervention, for an overall possible scoring range of 0-40. Higher scores associated with and increased level of patient fidelity. Overall scores will be summarized at each time point using basic descriptive statistics.
Change in Mood States (Quality of Life) | Baseline, 1 month post-operatively, 2 month post-operatively
  Change in mood states will be assessed using the Profile of Mood States (POMS) Inventory-Short form. POMS is an 11-item checklist of mood states which assesses psychological distress including tension, depression, and fatigue. The questionnaire consists of a list of adjectives and asks patients to provide a score best describing feelings associated with each particular adjective (mood state) over the past week based on a 5 point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely"), yielding an overall possible scoring range of 0-44. Overall scores will be summarized at each time point using basic descriptive statistics. Higher scores are associated with an increased level of distress and negative mood states (including tension, depression, fatigue).

SECONDARY OUTCOMES:
Stressful Life Events | Baseline, 1 month post-operatively, 2 month post-operatively
  Stressful life events will be assessed using the List of Threatening Experiences - Questionnaire (LTE-Q). The LTE-Q is a 12-item survey used to assess acute stressful events that could influence quality of life and cortisol outcomes. Patients are provided with 12 questions and asked to provide a binary (Yes/No) response as to whether each event was experienced over the prior 12 month period. "No" responses are assigned a value of 0 and "Yes" responses are assigned a value of 1. Item scores are summed to derive a total score with an overall possible scoring range of 0-12. Overall scores will be summarized at each time point using basic descriptive statistics. Higher scores are associated with an increase in stressful life events and a negative impact on quality of life.
Religiosity | Baseline
  Religiosity will be assessed using the Duke University Religion Index (DUREL). The DUREL is 5-item survey that measures religious involvement in terms of public religious behavior (church activities), private behavior (praying), and intrinsic religiousness (involvement of religion in dealings in life). The first two statements ask patients about engagement with public and private religious meetings, respectively, and are scored on a scale of "1" (more than once/week; more than once/day, respectively) through "6" (never; rarely or never, respectively) based on frequency of engagement. The last three statements ask about religious beliefs/experiences based on a 5 point scale ranging from 1 ("Definitely true of me") to 5 ("Definitely not true"). Scores for the 5 statements are added for a possible overall range of 5-27. Overall scores will be summarized at each time point using basic descriptive statistics. Lower scores are associated with increased levels of religious involvement.
Spirituality | Baseline, 1 month post-operatively, 2 month post-operatively
  Spirituality will be assessed using the Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12). The FACIT-Sp-12 is a 12-item questionnaire which consists of statements which serve as a measure of spirituality that measures domains of meaning, peace, and faith. Patients are provided with 12 statements that people with similar illnesses have said are important and asked to provide a score indicating how true the particular statement is for them over the past 7 days, based on a 5 point Likert scale ranging from 0 ("Not at all") to 4 ("Extremely") for an overall range of 0-48. Overall scores will be summarized at each time point using basic descriptive statistics. Higher scores are associated with an increased level of spiritual well-being.
Pain Inventory (Quality of Life) | Baseline, 1 month post-operatively, 2 month post-operatively
  Pain Severity and Pain Interference will be assessed using the Brief Pain Inventory Short Form (BPI-SF). BPI-SF consists of statements that assess the severity of pain and its impact on functioning in patients with chronic illnesses. The BPI-SF uses a 0-10 numeric rating scale for item rating for 2 subscales: Pain Severity (4 items) and Pain Interference (7 items). Patients provide a Pain Severity score between 0 ("No Pain") and 10 ("Pain as bad as you can imagine") and a mean of the 4 severity items on the BPI-SF is determined. Similarly, patients are asked to provide a Pain Interference score between 0 ("Does not Interfere") and 10 ("Completely interferes") and a mean of the 7 interference items is determined. The two subscales are added for an overall possible range of 0-110. Overall scale scores will be summarized at each time point using basic descriptive statistics. Higher scores are associated with increased pain severity and an adverse impact on daily life function.
Cancer Behavior (Quality of Life) | Baseline, 1 month post-operatively, 2 month post-operatively
  Cancer behavior assessing four major constructs: maintaining independence; participating in medical care; coping and stress management; and managing affect, will be assessed using the Cancer Behavior Inventory Brief Form (CBI-B) form. The CBI-B survey consists of a 12-item scale which assesses how confident the patient is in performing specific behaviors during and after cancer treatment. Patients are asked to provide a score on a 9 point scale ranging from 1 ("Not at all Confident") to 9 ("Totally confident"), for an overall possible scoring range of 12-108. Overall scores will be summarized at each time point using basic descriptive statistics. Higher scores are associated with an increased level of self-efficacy in coping with cancer.
Blood Pressure | Baseline, 1 month post-operatively, 2 month post-operatively
  Blood pressure (BP) will be reported based on medical chart reviews. BP is comprised of a systolic pressure (arterial pressure during contraction) reading and a diastolic pressure (arterial pressure between heartbeats) reading, both measured in millimeters of mercury (mmHg), and reported as a single reading (systolic/diastolic). Optimal BP ranges can vary based on demographics however, in adults, elevated BP is a risk factor for adverse cardiovascular and cerebrovascular events. Group mean BP readings will be reported using basic descriptive statistics.
Heart Rate | Baseline, 1 month post-operatively, 2 month post-operatively
  Heart rate (HR) will be reported in beats per minute (BPM) at rest based on medical chart reviews. Target (resting) heart rate ranges can vary based on demographics however, in adults, a lower (resting) heart rate is correlated with a higher degree of fitness and a lower incidence of cardiovascular events. Group mean HR will be reported using basic descriptive statistics.
Respiration Rate | Baseline, 1 month post-operatively, 2 month post-operatively
  Respiration rate (RR) will be reported in breaths per minute (bpm) at rest based on medical chart reviews. Normal respiration rates for an adult can vary based on demographics but are generally 12-18 breaths per minute. Elevated respiration rates can be indicative of anxiety or other underlying health conditions. Group mean RR readings will be reported using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Moadel, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No